CLINICAL TRIAL: NCT00110045
Title: A Multicenter, Open, Phase II Study to Estimate the Activity and Safety of Caspofungin (CASP) in the First-Line Treatment of Probable and Proven Invasive Aspergillosis (IA) in Patients With Hematological Malignancies (HM) or Recipients of Autologous Haematopoietic Stem Cell Transplantation and Those With Allogeneic Haematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Caspofungin Acetate in Treating Aspergillosis in Patients With Hematologic Cancer or in Patients Who Have Undergone a Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Supportive Care
Other Study IDs: EORTC-65041; EORTC-65041; EUDRACT-2004-002944-90
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Cancer
Keywords: infection; ataxia-telangiectasia; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia in remission; recurrent adult T-cell leukemia/lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; prolymphocytic leukemia; recurrent adult Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; adult grade III lymphomatoid granulomatosis; recurrent adult grade III lymphomatoid granulomatosis; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; stage I grade 1 follicular lymphoma; stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; splenic marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; post-transplant lymphoproliferative disorder; extramedullary plasmacytoma; isolated plasmacytoma of bone; monoclonal gammopathy of undetermined significance; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; chronic myelomonocytic leukemia; disseminated neuroblastoma; high risk metastatic gestational trophoblastic tumor; recurrent neuroblastoma; recurrent ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; secondary acute myeloid leukemia; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; chronic phase chronic myelogenous leukemia; contiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; recurrent adult acute myeloid leukemia; stage I adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; T-cell large granular lymphocyte leukemia
MeSH Terms: conditions — Neoplasms; Infections; Ataxia Telangiectasia; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Neuroblastoma; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Breast Neoplasms; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Leukemia, Large Granular Lymphocytic | interventions — Caspofungin

INTERVENTIONS:
Drug: caspofungin acetate

SUMMARY:
RATIONALE: Antifungals, such as caspofungin acetate, may be effective in treating fungal infections caused by chemotherapy or stem cell transplant.

PURPOSE: This phase II trial is studying how well caspofungin acetate works as first-line treatment for aspergillosis in patients with hematologic cancer or in patients who have undergone a stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the activity of caspofungin acetate as first-line therapy for proven or probable invasive aspergillosis, in terms of response rate, in patients with hematologic malignancies or in patients who have undergone hematopoietic stem cell transplantation.

Secondary

* Determine the 84-day response rate in patients treated with this drug.
* Determine the 84-day survival rate in patients treated with this drug.
* Determine the safety of this drug, in terms of the rate of overall drug-related adverse events, the rate of overall drug-related serious adverse events, and the rate of drug-related adverse events leading to treatment discontinuation, in these patients.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to disease and/or type of prior hematopoietic stem cell transplantation (HSCT) (hematologic malignancy or autologous HSCT vs allogeneic HSCT).

Patients receive caspofungin acetate IV over approximately 1 hour once daily on days 1-15 in the absence of disease progression or unacceptable toxicity.

Patients achieving a complete response (CR) or partial response (PR) after day 15 may continue to receive caspofungin acetate as above until day 84 OR discontinue study treatment after day 15 and shift to an oral antifungal drug for maintenance therapy or prophylaxis, if considered to be in the best interest of the patient. Patients achieving stable disease after day 15 continue to receive caspofungin acetate as above until day 28. These patients then undergo a second evaluation. Patients who maintain stable disease continue to receive caspofungin acetate as above until day 84. Patients achieving CR or PR are treated as per CR or PR treatment described above.

After completion of study treatment, patients are followed weekly for 30 days.

PROJECTED ACCRUAL: A total of 149 patients (87 in stratum 1, 62 in stratum 2) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of proven or probable invasive aspergillosis (IA)

  * Patients with a diagnosis of possible IA are eligible provided they are upgraded to probable or proven IA by culture and/or histology results and Aspergillus galactomannan evaluation within 7 days after study entry
* Meets any of the following criteria:

  * Diagnosis of a hematologic malignancy
  * Underwent autologous or allogeneic hematopoietic stem cell transplantation

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 20-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* AST and ALT ≤ 5 times upper limit of normal (ULN)
* Bilirubin ≤ 5 times ULN
* Alkaline phosphatase ≤ 5 times ULN
* No severe hepatic insufficiency

  * Child-Pugh score ≤ 9

Renal

* No severe renal failure requiring hemodialysis or peritoneal dialysis
* Creatinine < 3.4 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception
* No known HIV positivity
* No history of allergy or adverse reaction to echinocandin drugs
* No known bacterial infection that is not adequately treated
* No psychological, familial, social, or geographical condition that would preclude study participation or compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Prior empirical antifungal therapy allowed provided treatment duration was ≤ 72 hours
* Prior prophylactic oral antifungals allowed
* Prior prophylactic IV fluconazole allowed
* More than 14 days since prior and no concurrent investigational agents
* No prior participation in this study
* No prior echinocandins
* No other concurrent antifungal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2005-02; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Response rate as assessed by standard criteria after completion of study treatment

SECONDARY OUTCOMES:
Response rate as assessed by standard and alternative criteria at 84 days and after completion of study treatment
Survival rate at 84 days
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Viscoli, MD, Study Chair — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (13):
- CHU Liege - Domaine Universitaire du Sart Tilman, Liège, Belgium
- France (4):
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Edouard Herriot - Lyon, Lyon
  - Hopital Saint-Louis, Paris
  - Hopital Universitaire Hautepierre, Strasbourg
- Medizinische Poliklinik, Universitaet Wuerzburg, Würzburg, Germany
- Italy (4):
  - Ospedale Santa Croce, Cuneo
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Ospedale San Martino, Genoa
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Hacettepe University - Faculty of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Viscoli C, Herbrecht R, Akan H, Baila L, Sonet A, Gallamini A, Giagounidis A, Marchetti O, Martino R, Meert L, Paesmans M, Ameye L, Shivaprakash M, Ullmann AJ, Maertens J; Infectious Disease Group of the EORTC. An EORTC Phase II study of caspofungin as first-line therapy of invasive aspergillosis in haematological patients. J Antimicrob Chemother. 2009 Dec;64(6):1274-81. doi: 10.1093/jac/dkp355. Epub 2009 Oct 19. PMID 19841031